CLINICAL TRIAL: NCT03007329
Title: A 24 Week Monocentric Prospective Randomized, Placebo-controlled Trial to Evaluate Efficacy of Combination of Exenatide and Dapagliflozin Compared to Dapagliflozin and Placebo and Its Effects on Hepatic, Myocardial and Pancreatic Fat Distribution in Patients With Uncontrolled Type 2 Diabetes Mellitus.
Brief Title: Effects of Combined Dapagliflozin and Exenatide Versus Dapagliflozin and Placebo on Ectopic Lipids in Patients With Uncontrolled Type 2 Diabetes Mellitus.
Acronym: EXENDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESR-15-10882
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Steatosis, Liver; Type2 Diabetes
Keywords: SGLT2 inhibitor; GLP1 agonist; type 2 Diabetes; steatosis of the liver; ectopic lipids; combined therapy
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus, Type 2 | interventions — Exenatide; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin & Exenatide (Active Comparator): Dapagliflozin 10mg orally once daily & Exenatide 2mg subcutaneous once weekly
  Interventions: Drug: Exenatide; Drug: Dapagliflozin
- Dapagliflozin & Placebo (Placebo Comparator): Dapagliflozin 10mg orally once daily & Exenatide matching Placebo 2mg subcutaneous once weekly
  Interventions: Drug: Exenatide matching Placebo; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Exenatide — Exenatide will be combined with Dapagliflozin
  Arms: Dapagliflozin & Exenatide
Drug: Exenatide matching Placebo — Exenatide matching Placebo will be combined with Dapagliflozin
  Arms: Dapagliflozin & Placebo
Drug: Dapagliflozin — Dapagliflozin, in both arms

SUMMARY:
SGLT2 antagonists and GLP1 agonists are used since a relatively short period as second line therapy if indicated and are well tolerated by patients featuring low risk of hypoglycaemia in comparison to insulin or other oral glucose lowering drug. This new treatment options offer an effective modality to lower blood glucose, if first line therapeutics fail. According to national and international guidelines combination of oral glucose lowering drugs is possible in multiple ways, but is currently not recommended for GLP1 agonists and SGLT2 inhibitors yet, as evidence and supporting studies are missing proving efficacy and safety]. Thus studies under standardized conditions are urgently needed to answer these unsolved questions.

First results of a combination of a SGLT2 Inhibitor and a GLP1 agonist demonstrated huge potential regarding glucose and weight reduction and safety issues. However, further studies are necessary to elucidate potential mechanisms of combination therapy with SGLT2 inhibitors and GLP1 agonists and its effect on weight loss, glucose control, effects on incretins and adipokines, as well as further effects on ectopic lipid accumulation in liver and other tissues as myocard or pancreas in humans.

As both monotherapies have effects on weight and metabolism, changes in abdominal, subcutaneous, hepatic, myocardial or pancreatic lipid content might be speculated and are focus of interest in this study. Recently GLP1 agonists were shown to have effects on hepatic lipid reduction in humans with diabetes.

Hepatic lipid content and steatosis hepatis are widely discussed to have major effects on progression of diabetes and cardiovascular disease. Thus reduction of lipid accumulation in hepatic tissue might have an effect on diabetes progression.

Also higher myocardial lipid accumulation is seen in diabetic patients probably partly responsible for higher cardiovascular risk in diabetics. So far results combining these two drug classes show less weight loss as might have been expected using monotherapy, so that further investigation will definitely shed light on combination of therapeutic concepts.

Facing a multiple of positive side effects (weight loss, blood pressure lowering, potential protective cardiac effects) using a combination of SGLT2 and GLP1 seems to be a promising therapeutic option in diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

T2DM

* Sex: male and female
* HbA1c >=6.5 and <=11
* Age >=18 and <=75 years
* BMI>=25kg/m2
* Metformin>=1000mg daily, 8 weeks stable dose Please note: Type 2 diabetes mellitus patients treated with less than 1000 mg metformin per day can only be included if the investigator considers the patient to be on the maximum tolerated dose and the investigator has documented the reason why uptitration to 1000 mg was not possible
* able and willing to not change diet and physical activity during enrollment in study
* consent and able to give informed consent.

Exclusion Criteria:

* other diabetes diagnosis than T2DM
* patients on other antidiabetic medication (Sulfonylurea, Glitazone, insulin for more than 2 weeks (see below), SGLT2 inhibitors, GLP1 agonist, nateglinide, repaglinide, acarbose, DPP4 inhibitors)
* Subjects currently or previously treated with insulin (with the exception of emergency situations in which insulin was given for less than 14 consecutive days, but not within the last 3 months before screening)
* known intolerance against study medication
* Contraindications including hypersensitivity known to metformin according to the local label
* recurrent urinary tract infections
* GFR < 60
* Liver enzymes above 3 fold normal range
* Bilirubin higher 3 fold normal range
* Any other clinical condition that would jeopardize patients safety while participating in this clinical trial
* disease at screening (other than NAFLD) such as relevant cardiovascular, gastrointestinal, hepatic, neurologic, psychiatric, endocrine (i.e. pancreatic) except T2DM, hematologic, malignant, infection or other major systemic diseases making implementation of the protocol or interpretation of the study results difficult
* history of pancreatitis
* Known autoimmune disease or chronic inflammatory condition
* Myocardial infarction or stroke within 6 months prior to screening
* Blood dyscrasias or any disorders causing haemolysis or unstable Red Blood Cell (e.g.malaria, babesiosis, haemolytic anaemia)
* Other liver disease including chronic viral hepatitis (B or C), alcohol abuse, hemochromatosis, alpha-1antitrypsin deficiency, autoimmune hepatitis, Wilson's disease, primary sclerosing cholangitis or primary biliary cirrhosis, or liver cirrhosis of any etiology
* malignancy within the last 5 years before randomisation
* medullary thyroid cancer
* family history of multiple endocrine neoplasia syndrome
* Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake
* Presence of any absolute or relative contraindication for the conduct of an MRI investigation, such as cardiac pacemakers, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators,cochlear implants, insulin pumps and nerve stimulators, prosthetic heart valves etc.
* History of bariatric surgery
* Treatment with anti-obesity drugs (e.g. sibutramine, orlistat) 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight
* Subjects receiving antihypertensive medication and/or thyroid hormones, the dose(s) of which have not been stable for at least 6 weeks prior to baseline
* Current treatment with systemic steroids at time of informed consent (Treatment with local and inhaled steroids is allowed)
* Use of drugs potentially associated with NAFLD for more than 2 consecutive weeks in the 6 months prior to screening.
* Use of anti-NASH drugs (thiazolidinediones, vitamin E, UDCA, SAM-e, betaine, milk thistle, anti-TNF therapies,) in the 3 months prior to randomization.
* Donation of blood (> 400 mL) during the previous 3 months prior to the screening visit or during the duration of the study
* Participation in another trial with an investigational drug within 30 days prior to informed consent.
* Any subject who is the investigator or any coinvestigator, research assistant, pharmacist, study coordinator, other staff thereof, directly involved in the conduct of the protocol.
* Pre-menopausal women (last menstruation ≤1 year prior to informed consent) who:
* are nursing or pregnant or
* are of child-bearing potential and are not practising an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives,sexual abstinence,( if acceptable by local authorities) double barrier method and vasectomised partner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
change in hepatic lipid content measured with magnetic resonance spectroscopy in % | baseline - week 24
  to investigate the effects on hepatic lipid content reduction of combination therapy with dapagliflozin (10mg daily) and exenatide (2mg weekly) compared to dapagliflozin (10mg daily) and placebo given for 24 weeks in patients with type 2 diabetes mellitus and insufficient glycaemic control despite oral therapy.

SECONDARY OUTCOMES:
change in myocardial lipid content measured with magnetic resonance spectroscopy in % | baseline - week 24
  to investigate the effects on myocardial lipid content reduction of combination therapy with dapagliflozin (10mg daily) and exenatide (2mg weekly) compared to dapagliflozin (10mg daily) and placebo given for 24 weeks in patients with type 2 diabetes mellitus and insufficient glycaemic control despite oral therapy.
change in pancreatic lipid content measured with magnetic resonance spectroscopy in % | baseline - week 24
  to investigate the effects on pancreatic lipid content reduction of combination therapy with dapagliflozin (10mg daily) and exenatide (2mg weekly) compared to dapagliflozin (10mg daily) and placebo given for 24 weeks in patients with type 2 diabetes mellitus and insufficient glycaemic control despite oral therapy.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | baseline- week 24
  safety and tolerability from baseline to end by number of participants with treatment related AEs and SAEs
Quality of Life questionnaire | baseline - week 24
  change from baseline in quality of live assessed by WHO Well Being Index
change in insulin resistance | baseline - week 24
  change from baseline in insulin resistance assessed by HOMA IR Index
change in insulin sensitivity | baseline - week 24
  change from baseline in insulin sensitivity assessed by OGIS
energy expenditure | baseline -week 24
  change from baseline of energy expenditure assessed by indirect calorimetry
energy intake | baseline -week 24
  change from baseline of energy intake assessed by 3 day eating protocols
blood pressure | baseline - week 24
  To assess the effect of combination therapy with dapagliflozin and exenatide on blood pressure compared to dapagliflozin and placebo.
weight loss | baseline - week 24.
  To assess the effect of combination therapy with dapagliflozin and exenatide on weight loss compared to dapagliflozin and placebo.
change in glomerular filtration rate | baseline -week 24
  change in GFR from baseline

OTHER OUTCOMES:
weight | baseline - week 24
  change in weight from baseline
hip circumference | baseline - week 24
  change in hip circumference from baseline
waist circumference | baseline - week 24
  change in waist circumference from baseline
fasting glucose | baseline - week 24
  change in fasting plasma glucose from baseline
HbA1c reduction >= 0.5% | baseline - week 24
  % of patient with HbA1c reduction of more than 0.5%
weight reduction >= 5% | baseline - week 24
  % of patient with weight reduction of more than 5%
change in triglycerides | baseline - week 24
  change in triglycerides from baseline
change in cholesterol | baseline - week 24
  change in cholesterol from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, Prof. Dr., Principal Investigator — Dep. of Medicine III, Div. of Endocrinology, Gender Medicine Unit
Locations (1):
- Abt. für Endokrinologie & Stoffwechsel, Univ. Klin f. Innere Medizin III, Vienna, Austria

REFERENCES:
- [Result] Harreiter J, Just I, Leutner M, Bastian M, Brath H, Schelkshorn C, Klepochova R, Krssak M, Kautzky-Willer A. Combined exenatide and dapagliflozin has no additive effects on reduction of hepatocellular lipids despite better glycaemic control in patients with type 2 diabetes mellitus treated with metformin: EXENDA, a 24-week, prospective, randomized, placebo-controlled pilot trial. Diabetes Obes Metab. 2021 May;23(5):1129-1139. doi: 10.1111/dom.14319. Epub 2021 Feb 10. PMID 33464703